CLINICAL TRIAL: NCT03830450
Title: Biomarkers in Estimation for Risk of Acute Kidney Injury in Cardiac Surgery
Brief Title: Biomarkers of Acute Kidney Injury in Cardiac Surgery
Acronym: AKIrisk
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nikola Bradic, MD (Other)
Responsible Party: Sponsor-Investigator, Nikola Bradic, MD, MD, Senior Lecturer, University Hospital Dubrava
Organization: University Hospital Dubrava (Other)
Other Study IDs: University North
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Acute Kidney Injury (Nontraumatic)
Keywords: Acute kidney injury; Cardiac surgery; NGAL; GDF-15
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute kidney injury (AKI) is the most common complication in patients after cardiac surgery. An usual estimation of risk for AKI is estimation of serum creatinine, which is unreliable indicator of AKI risk. Because of that, today different biomarkers are investigated to predict incidence for development AKI after cardiac surgery. This investigation will try to find potentially risk patients for developing AKI after cardiac surgery by using conventional markers (creatinine, glomerular filtration rate) in perioperative period comparing with two different biomarkers neutrophil gelatinase-associated lipocalin (NGAL) and growth differentiation factor 15 (GDF-15) which are proven markers in patients with increased risk for AKI development.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for cardiac surgery (CABG, valve replacement/repair, combined)
* older than 18 years

Exclusion Criteria:

* previous known renal disease
* patients on chronic dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cardiac surgery with usage of cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Consecutive values of neutrophil gelatinase-associated lipocalin (NGAL) | One year
  By the changing of NGAL values in consecutive measuring, predict which patients are in increased risk for development of AKI
Consecutive values of growth differentiation factor 15 (GDF-15) | One year
  By the changing of GDF-15 values in consecutive measuring, predict which patients are in increased risk for development of AKI
Consecutive values of glomerular filtration rate (GFR) | One Year
  By the changing of GFR values in consecutive measuring, predict which patients are in increased risk for development of AKI